CLINICAL TRIAL: NCT04920877
Title: APPLICATION OF NURSE-FOCUSED ALGORITHM IN INTENSIVE CARE UNITS TO PREVENT CENTRAL CATHETER-RELATED BLOODSTREAM İNFECTİONS
Brief Title: Preventing Central Catheter-Associated Bloodstream Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Aysun ACUN, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AIBU-SBF-AA-01
Record Dates: First submitted 2021-06-04; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Catheter Infection; Catheter Infections Related
Keywords: Catheter; Algorithms; Sepsis
MeSH Terms: conditions — Catheter-Related Infections; Sepsis

STUDY DESIGN:
Intervention Model Description: Patients followed with a central catheter in the intensive care unit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Central catheter-related bloodstream infection rates in intensive care units (Experimental)
  Interventions: Other: Infection Prevention

INTERVENTIONS:
Other: Infection Prevention — Preventing central catheter-related bloodstream infections in intensive care units

SUMMARY:
The research is an algorithm study focused on nursing care in order to prevent Central Catheter-Associated Bloodstream Infections in intensive care units. The algorithm prepared with infection control measures related to central catheter care will be applied with intensive care nurses and the effect of the algorithm on central catheter-related bloodstream infections will be examined. In practice, a 20-day preliminary assessment, a three-month intervention period, and a three-month post-intervention planning were made.

DETAILED DESCRIPTION:
In the light of literature review and guidelines, intensive care nurses will care for central catheters through an algorithm created with infection control measures.

Nurse-focused algorithm content to prevent central catheter-related bloodstream infections Hand hygiene practice Use of personal protective equipment according to infection control measures Evaluation of the catheter insertion site in terms of redness, swelling, tenderness, discharge, bleeding Use of >0.5% chlorhexidine solution containing 70% alcohol for skin antisepsis at the catheter insertion site (if there is no chlorhexidine, povidone iodine + 70% alcohol solution is used) Changing the transparent, semi-permeable dressings every 5-7 days and gauze dressings every 48 hours for catheter dressing Catheter dressing with aseptic technique Use of sterile, preservative-free saline for flushing and locking in order to ensure the lumen of the catheter.

Aseptic conditions should be observed if the junction of the catheter and the infusion set (Hub) is to be touched.

Keeping the used triple taps closed Changing IV fluid sets and connection tools at appropriate times Daily assessment of CVC requirement The research will be carried out in the 1st, 2nd and 3rd Level Intensive Care Units of Bilecik Training and Research Hospital in Bilecik, Turkey. Infection rates will be compared in the study. In the study, the date of June 2021 will be taken as a preliminary assessment and training time for nurses. July-September 2021 will be the intervention period of the study, and October-December 2021 will be the post-intervention period.

ELIGIBILITY:
Inclusion Criteria:

* A central venous catheter was inserted in the intensive care unit or before the intensive care unit admission, and being followed up in the intensive care unit with a central venous catheter.

Exclusion Criteria:

* Patients whose central venous catheter was terminated during intensive care follow-up.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06-04 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Infection rate | Three months
  Central catheter-related bloodstream infection rates in intensive care units

IPD SHARING:
Plan to Share IPD: No